CLINICAL TRIAL: NCT02856932
Title: Clinical Evaluation of Glass Ionomer With Glass Hybrid Technology Versus Conventional High Viscosity Glass Ionomer in Class I Cavities of High Caries Risk Patients: Randomized Controlled Trial
Brief Title: Clinical Evaluation of Glass Ionomer With Glass Hybrid Technology Versus Conventional High Viscosity Glass Ionomer in Class I Cavities of High Caries Risk Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Refaat El-Bialy, Assistant lecturer, Cairo University
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2016-08-178
Record Dates: First submitted 2016-08-01; First posted 2016-08-05 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Class I Cavities in High Caries Risk
MeSH Terms: interventions — glass ionomer

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Glass Ionomer with Glass Hybrid technology (Experimental): Intervention
  Interventions: Other: Glass ionomer with glass hybrid technology
- Conventional high viscosity Glass Ionomer (Active Comparator): Comparator
  Interventions: Other: Conventional high viscosity glass ionomer

INTERVENTIONS:
Other: Conventional high viscosity glass ionomer — Dental restorative material
  Other Names: GC EQUIA
  Arms: Conventional high viscosity Glass Ionomer
Other: Glass ionomer with glass hybrid technology — Dental restorative material
  Other Names: GC EQUIA Forte
  Arms: Glass Ionomer with Glass Hybrid technology

SUMMARY:
PICOTS:

P: High Caries Risk Patients with bilateral class I cavities. I: Glass Ionomer with Glass Hybrid Technology. C: Conventional High Viscosity Glass Ionomer. O: Clinical performance (Functional properties Biological properties) using (World Dental Federation) Fédération dentaire internationale (FDI) criteria for dental restorations.

T: 1 year. S: Randomized controlled Trial (split mouth design). Research question:In high caries risk patients with class I cavities will glass ionomer with glass hybrid technology has similar clinical performance as conventional high viscosity glass ionomer

ELIGIBILITY:
Inclusion Criteria:

* Bilateral class I carious lesions in their occlusal pits and fissures.
* High caries risk patients who has 1 or more cavitated lesion with risk factor declared by Caries Management By Risk Assessment (CAMBRA)
* Co-operative patients approving to participate in the trial.

Exclusion Criteria:

* Disabilities.
* Systemic diseases or severe medically compromised.
* Lack of compliance.
* Evidence of severe bruxism, clenching or temporomandibular joint disorders

Ages: 19 Years to 50 Years | Sex: All
Age Groups: Adult
Enrollment: 31 (Estimated)
Dates: Primary Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Clinical performance using FDI criteria for dental restorations (functional properties and biological properties) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of oral and dental medicine, cairo university, Cairo, Egypt